CLINICAL TRIAL: NCT01233050
Title: A Randomized Double-Blind Study of 2% Chlorhexidine Gluconate / 70% Isopropyl Alcohol vs Iodine Povacrylex [0.7% Available Iodine] / 74% Isopropyl Alcohol for Perioperative Skin Preparation in Open Elective Colorectal Surgery
Brief Title: Efficacy Comparison of Two Preoperative Skin Antisepsis Preparations in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EM-05-012087
Record Dates: First submitted 2010-10-22; First posted 2010-11-02 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Colorectal Surgery
Keywords: undergoing elective colon and /or rectal surgical procedures involving an abdominal incision
MeSH Terms: interventions — Ethanol; DuraPrep

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol (Active Comparator): Preoperative Skin Antisepsis Preparation
  Interventions: Drug: 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol
- Iodine Povacrylex/74% Isopropyl Alcohol (Active Comparator): Preoperative Skin Antisepsis Preparation
  Interventions: Drug: Iodine Povacrylex/74% Isopropyl Alcohol

INTERVENTIONS:
Drug: 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol — Preoperative skin antisepsis preparation
  Other Names: ChloraPrep
  Arms: 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol
Drug: Iodine Povacrylex/74% Isopropyl Alcohol — preoperative skin antisepsis preparation
  Other Names: DuraPrep
  Arms: Iodine Povacrylex/74% Isopropyl Alcohol

SUMMARY:
Surgical site infections (SSI) are one of the most common complications in the post-operative patient, and the second most common health care associated infection overall. It is estimated that there are between 500 thousand and 1.1 million surgical site infections in the United States each year. Given the magnitude of the problem, prevention of surgical site infections is a major goal of peri-operative care. However, skin preparation prior to surgery has not been as rigorously examined. The primary objective of this study is to compare the efficacy of two FDA approved, popular peri-operative skin preparations 2% chlorhexidine gluconate / 70% isopropyl alcohol to Iodine Povacrylex [0.7% available Iodine] / 74% Isopropyl Alcohol in the prevention of superficial surgical site infection. Male and female patients, age 18 years and older undergoing elective colorectal surgical procedures involving a laparotomy will be enrolled. These patients are at high risk of SSI. Eligible patients will be assessed at regular intervals for SSI and characterization of bacterial pathogen(s) in patients with SSI. Patients will remain enrolled into the study until 35 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older, male or female
2. Undergoing any large bowel procedure with an extraction incision site(including ileostomy closure and Hartman's colostomy reversals).
3. A clean-contaminated preoperative classification.
4. Patient must have decision-making capacity and undergo appropriate informed consent process.
5. Non-pregnant or post menopausal or surgically sterilized females. If of child-bearing age, patients must have a negative (serum or urine) pregnancy prior to surgery.

Exclusion Criteria:

1. Antibiotics taken within 5 days prior to surgery.
2. Infected wound classification.
3. Preoperative evaluation that may preclude full closure of the skin.
4. Undergoing any bowel procedure that will not result in an extraction incision.
5. Ongoing radiation or chemotherapy treatment.
6. Pregnant.
7. Refusal to accept medically indicated blood products.
8. Current abdominal wall infection or surgical site infection from previous laparotomy / laparoscopy.
9. History of laparotomy within the last 60 days.
10. Known allergy to iodine or to chlorhexidine gluconate.
11. Participating in a preoperative antibiotic trial.
12. Participating in a skin antisepsis trial.
13. Participating in Ulcerative colitis trial conflicting with this trial.
14. Women who are breast feeding (potential for transient hypothyroidism in the nursing newborn).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2010-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najjia N Mahmoud, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Broach RB, Paulson EC, Scott C, Mahmoud NN. Randomized Controlled Trial of Two Alcohol-based Preparations for Surgical Site Antisepsis in Colorectal Surgery. Ann Surg. 2017 Dec;266(6):946-951. doi: 10.1097/SLA.0000000000002189. PMID 28277409
- [Derived] Poulin P, Chapman K, McGahan L, Austen L, Schuler T. Preoperative skin antiseptics for preventing surgical site infections: what to do? ORNAC J. 2014 Sep;32(3):12-5, 24-9. PMID 25322531

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorhexidine-Alcohol: Preoperative Skin Antisepsis Preparation
  2% Chlorhexidine Gluconate/70% Isopropyl Alcohol: Preoperative skin antisepsis preparation
- Iodine Povacrylex-Alcohol: Preoperative Skin Antisepsis Preparation
  Iodine Povacrylex/74% Isopropyl Alcohol: preoperative skin antisepsis preparation
Period: Overall Study
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol
Started | 400 | 402
Completed | 392 (8 participants were excluded after treatment administered due to inclusion/exclusion criteria) | 396 (6 participants were excluded after treatment administered due to inclusion/exclusion criteria)
Not Completed | 8 | 6
Not completed — protocol deviation (inclusion/exclusion) | 8 | 6

BASELINE CHARACTERISTICS:
Population: Chlorhexidine-Alcohol arm - 8 participants were excluded after treatment administered due to inclusion/exclusion criteria
  Iodine Povacrylex-Alcohol Arm - 6 participants were excluded after treatment administered due to inclusion/exclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol | Total
Number analyzed (Participants) | 392 | 396 | 788
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.33 (16.65) | 56.75 (15.81) | 57.04 (16.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 203 | 405
  Male | 190 | 193 | 383
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 307 | 322 | 629
  African American or Black | 64 | 55 | 119
  Asian | 6 | 6 | 12
  Hispanic or Latino | 4 | 4 | 8
  Other | 1 | 3 | 4
  Unknown | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective Measures the Proportion of Patients With Superficial Site Infection as Defined by the CDC.
Description: The primary objective compares the efficacy of 2% chlorhexidine gluconate / 70% isopropyl alcohol (ChloraPrep) to Iodine Povacrylex [0.7% available Iodine] / 74% Isopropyl Alcohol (DuraPrep) in the prevention of superficial surgical site infection. The primary objective will be measured by the number and percentage of patients with superficial site infection as defined by the CDC.
Time Frame: within 35 days of randomization to treatment assignment
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol
Number analyzed (Participants) | 392 | 396
Participants | 40 | 46

2. Secondary Outcome: Time to Develop Surgical Site Infection
Description: average time from surgery to surgical site infection diagnosis
Time Frame: within 35 days of randomization to treatment assignment
Measure: Mean (Standard Error); unit: days
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol
Number analyzed (Participants) | 392 | 396
days | 8.0 (0.7) | 8.7 (0.6)

3. Secondary Outcome: Bacterial Pathogens Present in Documented Surgical Site Infection
Time Frame: within 35 days of randomization to treatment assignment
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol
Number analyzed (Participants) | 43 | 26
Participants | 43 | 26

4. Secondary Outcome: Number and Percentage of Participants With Deep Wound Infection
Time Frame: within 35 days of randomization to treatment assignment
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol
Number analyzed (Participants) | 392 | 396
Participants | 22 | 28

5. Secondary Outcome: Number and Percentage of Participants With Organ Space Infection
Time Frame: within 35 days of randomization to treatment assignment
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol
Number analyzed (Participants) | 392 | 396
Participants | 20 | 16

6. Secondary Outcome: Length of Hospital Stay
Time Frame: within 35 days of randomization to treatment assignment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol
Number analyzed (Participants) | 392 | 396
days | 7.0 (3.9) | 6.8 (3.7)

ADVERSE EVENTS:
Arm/Group | Chlorhexidine-Alcohol | Iodine Povacrylex-Alcohol
All-Cause Mortality (participants affected / at risk) | 1/392 | 1/396
Serious Adverse Events (participants affected / at risk) | 0/392 | 0/396
Other Adverse Events (participants affected / at risk) | 0/392 | 0/396

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No